CLINICAL TRIAL: NCT00325533
Title: Group Randomized Trial of a Barber-Based Intervention to Improve Hypertension Control in Black Men
Brief Title: Effectiveness of a Barbershop-Based Program to Improve High Blood Pressure Control and Awareness in Black Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Texas Southwestern Medical Center (Other); Donald W. Reynolds Foundation (Other)
Responsible Party: Ronald Victor, MD: Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 470; R01HL080582 (NIH); 55341; R01HL080582-01A2 (NIH)
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Blood Pressure, High; Blacks; African Americans
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening & Enhanced Intervention (Experimental): After an intensive 10-week baselne screening, the enhanced intervention group barbers will be trained to measure blood pressure and deliver health messages related to blood pressure control during each customer's visit.
  Interventions: Behavioral: Baseline BP Screening; Other: Intensive 10-week Blood Pressure Screening
- Screening (Active Comparator): After the intensive 10-week baseline BP screening (an intervention in itself), the barbershops in the comparison arm received a continual supply of American Heart Association pamphlets on Hypertension in African Americans.
  Interventions: Other: Intensive 10-week Blood Pressure Screening

INTERVENTIONS:
Behavioral: Baseline BP Screening — Barbers in the barbershops in the experimental arm will be trained to accurately measure and interpret blood pressure (BP). Each barber will offer a BP check to customers with each haircut, complete an encounter form after each haircut, discuss the BP reading with the customer, identify customers with elevated BP, and refer customers with elevated BP to a regular physician or other primary provider for long-term BP management. Each time a customer with elevated BP goes to a regular medical provider, he receives a free haircut, and the referring barber receives a monetary bonus.
  Arms: Screening & Enhanced Intervention
Other: Intensive 10-week Blood Pressure Screening — Intensive 10-week Blood Pressure Screening

SUMMARY:
Black men in the United States have a greater risk of developing high blood pressure than men of any other ethnic or racial group. The purpose of this study is to evaluate the effectiveness of a high blood pressure detection and medical referral program conducted by barbers in predominantly Black barbershops at increasing awareness and lowering blood pressure levels among their Black male customers.

DETAILED DESCRIPTION:
High blood pressure affects approximately 35% of Black men in the United States. This may be due to the fact that Black men frequently have an unusually high number of risk factors for high blood pressure, including diabetes, high stress levels, and increased salt intake and sensitivity. While high blood pressure can often be controlled through diet, lifestyle changes, or medication, it is a chronic asymptomatic medical condition for which individuals should remain under the care of a regular medical provider. A predominantly Black barbershop may be an optimum and receptive setting for an intervention that focuses on improving the detection and treatment of high blood pressure among Black men. In this study, barbers, deemed as influential peers, will be trained to continually monitor their customers' blood pressure, deliver health messages designed to change risk perception and ideas about healthcare utilization, and provide social support for changes in healthcare-seeking behavior and blood pressure levels. The purpose of this study is to evaluate the effectiveness of a barbershop-based intervention at increasing blood pressure awareness and lowering blood pressure levels among Black male customers. With over 18,000 Black barbershops in the United States, the results from this study may be extremely influential in improving the diagnosis and treatment of high blood pressure in Black men.

This study will enroll Black men who are regular customers at a participating barbershop. Each barbershop will be randomly assigned to either a 10-month intervention group or a control group. Nurses will train the intervention group barbers to measure blood pressure and deliver health messages related to blood pressure control during each customer's visit. Before and after the intervention, study researchers will interview barbers and customers over an 8-week period to collect information on blood pressure control. A 12-month follow-up visit will include assessments of blood pressure levels, customer recognition of elevated blood pressure levels, and the number of customers receiving regular medical care.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Regular customer at one of the participating barbershops

Exclusion Criteria:

* Does not speak English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2319 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percentage of customers with high blood pressure who achieve recommended systolic and diastolic blood pressure values | Measured at 12 months

SECONDARY OUTCOMES:
Customer recognition of elevated blood pressure levels | Measured at 12 months
Number of customers with high blood pressure with a regular medical provider | Measured at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Victor, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Rader F, Elashoff RM, Niknezhad S, Victor RG. Differential treatment of hypertension by primary care providers and hypertension specialists in a barber-based intervention trial to control hypertension in Black men. Am J Cardiol. 2013 Nov 1;112(9):1421-6. doi: 10.1016/j.amjcard.2013.07.004. Epub 2013 Aug 23. PMID 23978276
- [Derived] Victor RG, Ravenell JE, Freeman A, Leonard D, Bhat DG, Shafiq M, Knowles P, Storm JS, Adhikari E, Bibbins-Domingo K, Coxson PG, Pletcher MJ, Hannan P, Haley RW. Effectiveness of a barber-based intervention for improving hypertension control in black men: the BARBER-1 study: a cluster randomized trial. Arch Intern Med. 2011 Feb 28;171(4):342-50. doi: 10.1001/archinternmed.2010.390. Epub 2010 Oct 25. PMID 20975012
- [Derived] Victor RG, Ravenell JE, Freeman A, Bhat DG, Storm JS, Shafiq M, Knowles P, Hannan PJ, Haley R, Leonard D. A barber-based intervention for hypertension in African American men: design of a group randomized trial. Am Heart J. 2009 Jan;157(1):30-6. doi: 10.1016/j.ahj.2008.08.018. PMID 19081393